CLINICAL TRIAL: NCT00249353
Title: An Evaluation of the Safety and Effectiveness of CONCERTA® (Methylphenidate Hydrochloride), up to 72 mg Daily, in Adolescents With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: An Effectiveness and Safety Study of CONCERTA® (Methylphenidate Hydrochloride) in the Treatment of Adolescents With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002668
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Hyperactivity Disorder; ADHD; Concerta
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

INTERVENTIONS:
Drug: methylphenidate hydrochloride

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of CONCERTA® (methylphenidate hydrochloride, a central nervous system (CNS) stimulant) versus placebo for the treatment of Attention Deficit Hyperactivity Disorder (ADHD) in adolescents..

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety and effectiveness of CONCERTA® (methylphenidate hydrochloride) in the treatment of adolescents with Attention Deficit Hyperactivity Disorder (ADHD). This is a multicenter, randomized, double-blind, placebo-controlled study with adolescents ages 13-18 diagnosed with ADHD. The study consists of four phases. The Screening Phase establishes the diagnosis of ADHD and provides a one-week washout period without any ADHD medication. The Open-Label Titration Phase initiates the treatment of patients with one CONCERTA® 18 mg daily. Thereafter, the dose is increased approximately every 7 days in 18 mg increments (to a maximum of 72 mg daily), until an individualized dose is identified, based on the clinical judgment of the investigator. During the Double-Blind Phase, subjects are randomized to receive either their individualized CONCERTA® dose or a placebo, for a period of 2 weeks. Subjects who successfully complete the Double-Blind Phase are eligible to receive CONCERTA® for an 8-week, Open-Label, Follow-up Phase. The primary efficacy measurement is the total score of the ADHD Rating Scale, evaluated by the investigator at the end of the Double-Blind Phase. Safety assessments include monitoring adverse events, electrocardiograms (ECG), blood pressure, pulse, height and weight throughout the course of the study. The study hypothesis is that CONCERTA® is more effective than placebo in the treatment of Attention Deficit Hyperactivity Disorder in adolescents, and is well tolerated.

Titration Phase: CONCERTA® 18 mg taken orally, once daily, and increased approximately every 7 days in 18 mg increments up to a maximum daily dose of 72 mg. Double-Blind Phase: Individualized dose of CONCERTA® or placebo for 2 weeks. Open-Label Phase: Individualized dose of CONCERTA® for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Attention Deficit Hyperactivity Disorder (ADHD) as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV)
* Children's Global Assessment Scale rating of 41-70 at baseline (Screening Phase)

Exclusion Criteria:

* Subjects who are known to not respond to methylphenidate
* Have had adverse experiences from methylphenidate or hypersensitivity to CONCERTA or its components
* Have marked anxiety, tension or agitation
* Have glaucoma, ongoing seizure disorder, psychotic disorder, Tourette's disorder or family history of Tourette's disorder

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220 (Actual)
Dates: Start 2002-03; Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Total score on the Attention Deficit Hyperactivity Disorder (ADHD) Rating Scale, evaluated by the investigator at the end of the Double-Blind Phase.

SECONDARY OUTCOMES:
Attention Deficit Hyperactivity Disorder (ADHD) Rating Scale score, parent-evaluated weekly during Titration and Double-Blind Phases; Global Assessment of Effectiveness measured weekly during the Titration and Double-Blind Phases; Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.

REFERENCES:
- [Result] Wilens TE, McBurnett K, Bukstein O, McGough J, Greenhill L, Lerner M, Stein MA, Conners CK, Duby J, Newcorn J, Bailey CE, Kratochvil CJ, Coury D, Casat C, Denisco MJ, Halstead P, Bloom L, Zimmerman BA, Gu J, Cooper KM, Lynch JM. Multisite controlled study of OROS methylphenidate in the treatment of adolescents with attention-deficit/hyperactivity disorder. Arch Pediatr Adolesc Med. 2006 Jan;160(1):82-90. doi: 10.1001/archpedi.160.1.82. PMID 16389216
- [Derived] Newcorn JH, Stein MA, Cooper KM. Dose-response characteristics in adolescents with attention-deficit/hyperactivity disorder treated with OROS methylphenidate in a 4-week, open-label, dose-titration study. J Child Adolesc Psychopharmacol. 2010 Jun;20(3):187-96. doi: 10.1089/cap.2009.0102. PMID 20578931